CLINICAL TRIAL: NCT02881372
Title: Safety and Feasibility of Oral Food Desensitization in Children With Eosinophilic Esophagitis
Brief Title: EoE Food Desensitization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Tu Thanh Mai, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-17-0391
Record Dates: First submitted 2016-08-11; First posted 2016-08-29 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: oral food desensitization; food elimination; food reintroduction
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral food desensitization (Experimental): All of the children enrolled in the study will receive oral food desensitization with his or her specific EoE flare-inducing food antigen (e.g. cow's milk protein). The food antigen will be diluted in a 50% glycerin/water solution containing ascorbic acid (Vitamin C) to stabilize and preserve the solution. This oral spray will need to be administered twice a day, every day for a total of 4 months.
  Interventions: Other: Oral food desensitization

INTERVENTIONS:
Other: Oral food desensitization — The child's specific food antigen will be diluted in a 50% glycerin/water solution containing ascorbic acid (Vitamin C). This oral spray solution will need to be administered twice a day, every day for a total of 4 months

SUMMARY:
This is a single-center, prospective, pilot clinical trial in which children ages 3-17 years with eosinophilic esophagitis (EoE) who have a known food that triggers EoE flares receive oral desensitization with that specific food antigen, followed by reintroduction of that food into the diet. The purpose of this study is to investigate the safety and feasibility of oral desensitization in children with EoE so that, if determined to be safe, can be repeated on a larger scale to determine efficacy.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a clinicopathologic disorder of the esophagus triggered by food and/or environmental allergens and is characterized by symptoms of esophageal dysfunction and eosinophilia of the esophagus. Current therapy is centered on controlling inflammation with steroids and/or food antigen avoidance. Such treatment options have significant side effects and reduce quality of life, especially in children. The purpose of the study is to discover a way for flare-provoking foods to be reintroduced into the child's diet without the need for medical therapy.

The study would involve children ages 3-17 years with biopsy-proven EoE who have a known flare-inducing food trigger. Following baseline blood work and esophagogastroduodenoscopy (EGD), the investigators will initiate oral desensitization treatment in which the child swallows a spray solution containing his or her specific food allergen extract in increasing concentrations twice daily for 4 months. The next phase of the study would involve reintroduction of the actual food for 4 weeks followed by repeat blood work and EGD. Success would be defined by having a peak eosinophil count <15 per high power field on the final esophageal biopsy.

Oral food desensitization has been well-studied in patients with food allergies but never in patients with pre-existing EoE. In those studies, the adverse events included mild reactions, such as watery eyes, rhinitis, sneezing, throat pruritus, transient erythema and abdominal pain. These reactions usually did not require stopping desensitization and were well controlled by antihistamines and steroids. Benefits include children having a less restricted diet and eliminating the need for steroid therapy. This study should yield valuable information regarding the management of EoE, thereby improving the current understanding of its pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patient, ages 3-17 years, with known diagnosis of EoE based upon esophageal biopsy demonstrating ≥15 eos/hpf and lack of symptomatic or histological response to PPI therapy and/or normal esophageal pH evaluation.
2. Known or suspected flare-inducing food trigger based upon supporting histological evidence.
3. Already undergoing a baseline EGD followed by food reintroduction and repeat EGD, as standard of care at the recommendation of the child's gastroenterologist.
4. Signed informed consent for the subject's participation in the study provided by the parent/ legal guardian and child/adolescent assent for subjects 7-17 years.
5. Assent by the patient's pediatric gastroenterologist for the patient's participation in the study.

Exclusion Criteria:

1. Presence of other disorders associated with similar clinical, histological or endoscopic features, such as PPI-responsive esophageal eosinophilia, esophageal eosinophilia associated with gastroesophageal reflux disease (GERD), Crohn's disease, infectious esophagitis (i.e. herpes simplex virus or candida), drug-associated esophagitis, collagen vascular disease, hypereosinophilic syndrome and eosinophilic gastroenteritis.
2. Previous or current diagnosis of cancer or leukemia.
3. History of chemotherapy within the past 3 months.
4. History of esophageal stricture or food impaction.
5. History of anaphylaxis or other severe adverse reaction to the specific food trigger being tested.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Peak eosinophil count on esophageal biopsy | 5 months
  Remission of esophageal eosinophilia as defined by having <15 eosinophils per high power field on peak esophageal biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rhoads, MD, Study Director — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Gupta SK. Noninvasive markers of eosinophilic esophagitis. Gastrointest Endosc Clin N Am. 2008 Jan;18(1):157-67; xi. doi: 10.1016/j.giec.2007.09.004. PMID 18061109
- [Background] Arias A, Perez-Martinez I, Tenias JM, Lucendo AJ. Systematic review with meta-analysis: the incidence and prevalence of eosinophilic oesophagitis in children and adults in population-based studies. Aliment Pharmacol Ther. 2016 Jan;43(1):3-15. doi: 10.1111/apt.13441. Epub 2015 Oct 28. PMID 26510832
- [Background] Dellon ES, Gonsalves N, Hirano I, Furuta GT, Liacouras CA, Katzka DA; American College of Gastroenterology. ACG clinical guideline: Evidenced based approach to the diagnosis and management of esophageal eosinophilia and eosinophilic esophagitis (EoE). Am J Gastroenterol. 2013 May;108(5):679-92; quiz 693. doi: 10.1038/ajg.2013.71. Epub 2013 Apr 9. PMID 23567357
- [Background] Cianferoni A, Spergel JM. Immunotherapeutic approaches for the treatment of eosinophilic esophagitis. Immunotherapy. 2014;6(3):321-31. doi: 10.2217/imt.14.3. PMID 24762076
- [Background] Simon D, Cianferoni A, Spergel JM, Aceves S, Holbreich M, Venter C, Rothenberg ME, Terreehorst I, Muraro A, Lucendo AJ, Schoepfer A, Straumann A, Simon HU. Eosinophilic esophagitis is characterized by a non-IgE-mediated food hypersensitivity. Allergy. 2016 May;71(5):611-20. doi: 10.1111/all.12846. Epub 2016 Feb 25. PMID 26799684
- [Background] Schlag C, Miehlke S, Heiseke A, Brockow K, Krug A, von Arnim U, Straumann A, Vieth M, Bussmann C, Mueller R, Greinwald R, Bajbouj M. Peripheral blood eosinophils and other non-invasive biomarkers can monitor treatment response in eosinophilic oesophagitis. Aliment Pharmacol Ther. 2015 Nov;42(9):1122-30. doi: 10.1111/apt.13386. Epub 2015 Aug 27. PMID 26314389
- [Background] Kagalwalla AF, Shah A, Li BU, Sentongo TA, Ritz S, Manuel-Rubio M, Jacques K, Wang D, Melin-Aldana H, Nelson SP. Identification of specific foods responsible for inflammation in children with eosinophilic esophagitis successfully treated with empiric elimination diet. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):145-9. doi: 10.1097/MPG.0b013e31821cf503. PMID 21788754
- [Background] Molina-Infante J, Arias A, Barrio J, Rodriguez-Sanchez J, Sanchez-Cazalilla M, Lucendo AJ. Four-food group elimination diet for adult eosinophilic esophagitis: A prospective multicenter study. J Allergy Clin Immunol. 2014 Nov;134(5):1093-9.e1. doi: 10.1016/j.jaci.2014.07.023. Epub 2014 Aug 28. PMID 25174868
- [Background] Spergel JM, Shuker M. Nutritional management of eosinophilic esophagitis. Gastrointest Endosc Clin N Am. 2008 Jan;18(1):179-94; xi. doi: 10.1016/j.giec.2007.09.008. PMID 18061111
- [Background] Pajno GB, Cox L, Caminiti L, Ramistella V, Crisafulli G. Oral Immunotherapy for Treatment of Immunoglobulin E-Mediated Food Allergy: The Transition to Clinical Practice. Pediatr Allergy Immunol Pulmonol. 2014 Jun 1;27(2):42-50. doi: 10.1089/ped.2014.0332. PMID 24963452
- [Background] Howie SR. Blood sample volumes in child health research: review of safe limits. Bull World Health Organ. 2011 Jan 1;89(1):46-53. doi: 10.2471/BLT.10.080010. Epub 2010 Sep 10. PMID 21346890
- [Background] Martin LJ, Franciosi JP, Collins MH, Abonia JP, Lee JJ, Hommel KA, Varni JW, Grotjan JT, Eby M, He H, Marsolo K, Putnam PE, Garza JM, Kaul A, Wen T, Rothenberg ME. Pediatric Eosinophilic Esophagitis Symptom Scores (PEESS v2.0) identify histologic and molecular correlates of the key clinical features of disease. J Allergy Clin Immunol. 2015 Jun;135(6):1519-28.e8. doi: 10.1016/j.jaci.2015.03.004. PMID 26051952
- [Background] Franciosi JP, Hommel KA, DeBrosse CW, Greenberg AB, Greenler AJ, Abonia JP, Rothenberg ME, Varni JW. Development of a validated patient-reported symptom metric for pediatric eosinophilic esophagitis: qualitative methods. BMC Gastroenterol. 2011 Nov 18;11:126. doi: 10.1186/1471-230X-11-126. PMID 22099448
- [Background] Peters RL, Dang TD, Allen KJ. Specific oral tolerance induction in childhood. Pediatr Allergy Immunol. 2016 Dec;27(8):784-794. doi: 10.1111/pai.12620. Epub 2016 Sep 16. PMID 27496561
- [Background] Spergel JM, Brown-Whitehorn TF, Beausoleil JL, Franciosi J, Shuker M, Verma R, Liacouras CA. 14 years of eosinophilic esophagitis: clinical features and prognosis. J Pediatr Gastroenterol Nutr. 2009 Jan;48(1):30-6. doi: 10.1097/MPG.0b013e3181788282. PMID 19172120
- [Background] Lucendo AJ, Sanchez-Cazalilla M. Adult versus pediatric eosinophilic esophagitis: important differences and similarities for the clinician to understand. Expert Rev Clin Immunol. 2012 Nov;8(8):733-45. doi: 10.1586/eci.12.68. PMID 23167685
- See also: Select Committee on GRAS Substances (SCOGS) Opinion: L-ascorbic acid, sodium L-ascorbate, calcium L-ascorbate, ascorbyl palmitate (palmitoyl L-ascorbic), erythorbic acid (D-isoascorbic acid), and sodium erythorbate (sodium D-isoascorbate) — http://wayback.archive-it.org/7993/20180123233947/https:/www.fda.gov/Food/IngredientsPackagingLabeling/GRAS/SCOGS/ucm260452.htm